CLINICAL TRIAL: NCT05181124
Title: Clinical Trial To Evaluate Pharmacokinetic Interactions and Safety Between JP-1366 and Aceclofenac, Meloxicam, and Naproxen in Korean Healthy Volunteers and Compare Pharmacokinetics and Safety of JP-1366 Between Korean and Caucasian
Brief Title: Compare Pharmacokinetics and Safety of JP-1366 Between Korean and Caucasian
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: JP-1366-103
Record Dates: First submitted 2021-11-23; First posted 2022-01-06 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-01

CONDITIONS: Anti-Ulcer Agents
MeSH Terms: interventions — aceclofenac; Meloxicam; Naproxen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- JP-1366 and aceclofenac (Experimental)
  Interventions: Drug: coadministration of JP-1366 and aceclofenac
- JP-1366 and meloxicam (Experimental)
  Interventions: Drug: coadministration of JP-1366 and meloxicam
- JP-1366 and naproxen (Experimental)
  Interventions: Drug: coadministration of JP-1366 and naproxen
- JP-1366 (Experimental)
  Interventions: Drug: single-dosing of JP-1366 in Korean and Caucasian

INTERVENTIONS:
Drug: coadministration of JP-1366 and aceclofenac — An open-label, multiple-dosing, fixed sequence, 3-period design
  Arms: JP-1366 and aceclofenac
Drug: coadministration of JP-1366 and meloxicam — An open-label, multiple-dosing, fixed sequence, 3-period design
  Arms: JP-1366 and meloxicam
Drug: coadministration of JP-1366 and naproxen — An open-label, multiple-dosing, fixed sequence, 3-period design
  Arms: JP-1366 and naproxen
Drug: single-dosing of JP-1366 in Korean and Caucasian — An open-label, single-dosing, parallel design
  Arms: JP-1366

SUMMARY:
To evaluate the effect of coadministration of aceclofenac, meloxicam and naproxen on pharmacokinetic interactions and safety of JP-1366 in healthy Korean subjects and to compare the pharmacokinetic nature and safety of JP-1366 between healthy Korean and Caucasian.

ELIGIBILITY:
Inclusion Criteria:

* Subject who has fully informed about this study and understand co mpletely, decide to participate voluntarily and agree with the writte n consent before screening test.
* A healthy volunteer in the age of upper 19 at the time of the scree ning test.
* Subject whose BMI was 18.0 or more and 30.0 or less and whose b ody weight was 50kg or more if in male, and 45kg or more if in fe male at the same time.
* Caucasian in Part 4 who has medical interview and documents(passport, birth certificate) or signatured conformation by the subject.

Exclusion Criteria:

* The Subject who has clinically significant diseases with liver, kidney, nervous system, digestive system, immune system, respiratory system, and endocrine system, musculoskeletal system or the blood or tumor disease, cardiovascular disease (including orthostatic hypotension), mental disorder or with history of the disease.
* The subject who has a history of gastrointestinal disorders (gastrointestinal ulcers, gastritis, gastric ulcer, gastroesophageal reflux disease, Crohn's disease, etc.) or history of gastrointestinal surgery that may affect the safety and PK/PD Evaluation of the investigational product (Except for simple cecal surgery and hernia surgery)
* The subject who has a hereditary disorder (galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption etc.).
* The subject who has a history of an active peptic ulcer or bleeding.
* Screening laboratory test showing any of the following abnormal laboratory results: ALT, AST, Total bilirubin > 2.0 x ULN - e-GFR < 60 mL/min/1.73m2 (CKD-EPI formula) - Positive result for Serological test (HBsAg, HCV Ab, HIV Ab, Syphilis regain test)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Part 1 | Single dosing of aceclofenac: 1day 0hour (before IP administration), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12hour
  - Cmax,ss of JP-1366
Part 1 | Single dosing of aceclofenac: 1day 0hour (before IP administration), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12hour
  - AUCτ,ss of JP-1366
Part 1 | Single dosing of aceclofenac: 1day 0hour (before IP administration), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12hour
  - Cmax aceclofenac
Part 1 | Single dosing of aceclofenac: 1day 0hour (before IP administration), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12hour
  - AUCτ aceclofenac
Part 1 | Single dosing of JP-1366: 4day 0hour, 6day 0hour, 7day 0hour, 8day 0hour (before IP administration), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24hour (9day 0hour)
  - Cmax,ss of JP-1366
Part 1 | Single dosing of JP-1366: 4day 0hour, 6day 0hour, 7day 0hour, 8day 0hour (before IP administration), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24hour (9day 0hour)
  - AUCτ,ss of JP-1366
Part 1 | Single dosing of JP-1366: 4day 0hour, 6day 0hour, 7day 0hour, 8day 0hour (before IP administration), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24h (9day 0hour)
  - AUCτ of aceclofenac
Part 1 | Single dosing of JP-1366: 4day 0hour, 6day 0hour, 7day 0hour, 8day 0hour (before IP administration), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24hour (9day 0hour)
  - Cmax of aceclofenac
Part 1 | Coadministration of JP-1366 and aceclofenac: 9day 0hour (before IP administration), 0.25, 0.5, 0.75† , 1, 1.5, 2, 2.5‡ , 3, 4, 6, 8, 10, 12, 24hour (10day 0hour)
  - Cmax,ss of JP-1366
Part 1 | Coadministration of JP-1366 and aceclofenac: 9day 0hour (before IP administration), 0.25, 0.5, 0.75† , 1, 1.5, 2, 2.5‡ , 3, 4, 6, 8, 10, 12, 24hour (10day 0hour)
  - AUCτ,ss of JP-1366
Part 1 | Coadministration of JP-1366 and aceclofenac: 9day 0hour (before IP administration), 0.25, 0.5, 0.75† , 1, 1.5, 2, 2.5‡ , 3, 4, 6, 8, 10, 12, 24hour (10day 0hour)
  - Cmax of aceclofenac
Part 1 | Coadministration of JP-1366 and aceclofenac: 9day 0hour (before IP administration), 0.25, 0.5, 0.75† , 1, 1.5, 2, 2.5‡ , 3, 4, 6, 8, 10, 12, 24hour (10day 0hour)
  - AUCτ of aceclofenac
Part 2 | Single dosing of JP-1366: 1day 0hour, 3day 0hour, 4day 0hour, 5day 0hour (before IP administration), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24hour (6day 0hour), 15day 0hour (before IP administration)
  - Cmax,ss of JP-1366, meloxicam
Part 2 | Single dosing of JP-1366: 1day 0hour, 3day 0hour, 4day 0hour, 5day 0hour (before IP administration), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24hour (6day 0hour), 15day 0hour (before IP administration)
  - AUCτ,ss of JP-1366, meloxicam
Part 2 | Single dosing of Meloxicam: 19day 0hour (before IP administration), 1, 2, 3, 4, 5, 6, 8, 12, 24hour (20day 0hour)
  - Cmax,ss of JP-1366, meloxicam
Part 2 | Single dosing of Meloxicam: 19day 0hour (before IP administration), 1, 2, 3, 4, 5, 6, 8, 12, 24hour (20day 0hour)
  - AUCτ,ss of JP-1366, meloxicam
Part 2 | Coadministration of JP-1366 and meloxicam: 22day 0hour† , 24day 0hour† , 25day 0hour† , 26day 0hour (before IP administration), 0.25† , 0.5† , 0.75† , 1, 1.5† , 2, 3, 4, 5‡ , 6, 8, 10† , 12, 24hour (27day 0hour)
  - Cmax,ss of JP-1366, meloxicam
Part 2 | Coadministration of JP-1366 and meloxicam: 22day 0hour† , 24day 0hour† , 25day 0hour† , 26day 0hour (before IP administration), 0.25† , 0.5† , 0.75† , 1, 1.5† , 2, 3, 4, 5‡ , 6, 8, 10† , 12, 24hour (27day 0hour)
  - AUCτ,ss of JP-1366, meloxicam
Part 3 | Single dosing of JP-1366: 1day 0hour, 3day 0hour, 4day 0hour, 5day 0hour (before IP administration), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24hour (6day 0hour), 15day 0hour (before IP administration)
  - Cmax,ss of JP-1366, naproxen
Part 3 | Single dosing of JP-1366: 1day 0hour, 3day 0hour, 4day 0hour, 5day 0hour (before IP administration), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24hour (6day 0hour), 15day 0hour (before IP administration)
  - AUCτ,ss of JP-1366, naproxen
Part 3 | Single dosing of naproxen: 19day 0hour (before IP administration), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12hour
  - Cmax,ss of JP-1366, naproxen
Part 3 | Single dosing of naproxen: 19day 0hour (before IP administration), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12hour
  - AUCτ,ss of JP-1366, naproxen
Part 3 | Coadministration of JP-1366 and naproxen: 22day 0hour† , 24day 0hour† , 25day 0hour† , 26day 0hour (before IP administration), 0.25† , 0.5, 0.75† , 1, 1.5, 2, 2.5‡ , 3, 4, 5, 6, 8, 10† , 12, 24hour (27day 0hour)
  - Cmax,ss of JP-1366, naproxen
Part 3 | Coadministration of JP-1366 and naproxen: 22day 0hour† , 24day 0hour† , 25day 0hour† , 26day 0hour (before IP administration), 0.25† , 0.5, 0.75† , 1, 1.5, 2, 2.5‡ , 3, 4, 5, 6, 8, 10† , 12, 24hour (27day 0hour)
  - AUCτ,ss of JP-1366, naproxen
Part 4 | 1day 0hour (before IP administration), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 (2day 0hour), 48hour (3day 0hour)
  - Cmax of JP-1366 in Korean and Caucasian
Part 4 | 1day 0hour (before IP administration), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 (2day 0hour), 48hour (3day 0hour)
  - AUClast of JP-1366 in Korean and Caucasian

CONTACTS AND LOCATIONS:
Locations (1):
- Cha University Bundang Medical Center, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No